CLINICAL TRIAL: NCT04554797
Title: Regional Hypothermia in Combination With Endovascular Thrombectomy in Acute Ischemic Stroke
Acronym: RE-HIBER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RE-HIBER
Record Dates: First submitted 2020-09-13; First posted 2020-09-18 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Stroke; Neuroprotection; Hypothermia
MeSH Terms: conditions — Stroke; Hypothermia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regional Hypothermia group (Experimental)
  Interventions: Other: Regional Hypothermia
- Control group (No Intervention)

INTERVENTIONS:
Other: Regional Hypothermia — Regional hypothermia was achieved by intraarteral perfusion of cold fluid into the ischemic area of the brain
  Arms: Regional Hypothermia group

SUMMARY:
The investigators have previous shown that regional hypothermia by the intra-arterial infusion of cold saline combined with mechanical thrombectomy in acute ischemic stroke is feasible and safe. The safety of selective brain cooling in patients undergoing mechanical thrombectomy, however, is not established in a randomized trial. The investigators therefore conducted this RCT study to further explore the safety of regional hypothermia in patients with acute ischemic stroke who underwent mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤80
* Clinical signs consistent with the diagnosis of an acute ischemic stroke
* Baseline NIHSS score obtained prior to randomization ≥8
* Intracranial arterial occlusion of the distal intracranial carotid artery or
* Middle (M1/M2), demonstrated with CTA, MRA, DSA
* The possibility to start treatment (artery puncture) within 6 hours from onset
* Regional hypothermia is expected to start within 15 minutes after recanalization
* Informed consent given

Exclusion Criteria:

* mTICI<2b after endovascular treatment
* No significant pre-stroke disability (mRS ≤1)
* Previous NYHA grade > 1
* Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 3.0
* Baseline platelet count < 50000/µL
* Baseline blood glucose of < 50mg/dL or >400mg/dl
* Severe, sustained hypertension (SBP > 220 mm Hg or DBP > 110 mm Hg). NOTE: If the blood pressure can be successfully reduced and maintained at the acceptable level using local treatment guidelines recommended medication (including iv antihypertensive drips), the patient can be enrolled.
* Seizures at stroke onset which would preclude obtaining a baseline NIHSS
* Subjects who have received iv t-PA treatment beyond 4,5 hours from the beginning of the symptoms
* Renal insufficiency with creatinine ≥ 3 mg/dl
* Woman of childbearing potential who is known to be pregnant or lactating
* Subject participating in a study involving an investigational drug or device that would impact this study
* Cerebral vasculitis
* Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations
* Unlikely to be available for 3 months follow-up (e.g. no fixed home address, visitor from overseas).
* CT or MR evidence of hemorrhage (the presence of microbleeds on MRI is allowed)
* ASPECT<6
* Subjects with occlusions in multiple vascular territories (anterior circulation and posterior circulation)
* Evidence of intracranial tumor (except small meningioma)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-16 (Estimated); Primary Completion 2020-12-16 (Estimated); Study Completion 2021-03-16 (Estimated)

PRIMARY OUTCOMES:
Rate of any major adverse events | 7 days

SECONDARY OUTCOMES:
Rate of intracerebral hemorrhage | 24 hours
Rate of symptomatic intracerebral hemorrhage | 24 hours
Rate of death | 90 days
NIHSS | 24 hours
  Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating more severe neurologic deficits.
Final infarct volume | 5-7 days
  measured on 5-7 days CT (or MRI if available)
NIHSS | 7 days or discharge
  Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating more severe neurologic deficits.
Modified Rankin scale | 90 days
  The modified Rankin scale is a 7-point scale ranging from 0 (no symptoms) to 6 (death). A score of 2 or less indicates functional independence.

OTHER OUTCOMES:
Rate of vessel recanalization after treatment | 24 hours
  Assessed by CTA or MRA
The temperature change of the tympanic membrane on the ipsilateral side of the vascular occlusion within one hour after endovascular treatment | 1 hour
The patient's rectal temperature within one hour after endovascular treatment | 1 hour

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Lu He hospital, Capital Medical University, Beijing, Beijing Municipality